CLINICAL TRIAL: NCT04382235
Title: Management Through Non-invasive Ventilatory Support of Patients Showing an Acute Respiratory Failure Related to COVID-19 in Non-intensive Wards
Brief Title: Non-invasive Ventilatory Support of Patients Affected by COVID-19
Acronym: WARd-COVID
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: WARd-COVID
Record Dates: First submitted 2020-05-05; First posted 2020-05-11 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2021-04

CONDITIONS: Covid-19
Keywords: Coronavirus; sars-covid-2; coronavirus infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Noninvasive Ventilation; Continuous Positive Airway Pressure; Head Protective Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid-19 related Pneumonia patients: The cohort is defined by subjects with a diagnosis of COVID 19-related pneumonia requiring non-invasive ventilatory support.
  Interventions: Device: Non-invasive ventilatory support

INTERVENTIONS:
Device: Non-invasive ventilatory support — All non-invasive ventilatory support wll be recorded. All collected data is taken and monitored during normal clinical practice without adding any other tests.
  Other Names: High-flow nasal cannulas (HFNC); Non-invasive ventilation (NIV); Continuous positive airway pressure (CPAP) delivered with a face mask or helmet (helmet)

SUMMARY:
Prospective, observational, multicenter study aiming to evaluate the number of COVID-19 pneumonia related patients treated with non-invasive ventilatory support outside the intensive care unit.

In addition, the study aims to obtain information related to the clinical characteristics and hospital results of these patients.

DETAILED DESCRIPTION:
In February 2020, the first case of transmission of the syndrome, indicated as COVID-19, was reported in Italy. Unfortunately, during March 2020, the syndrome spread rapidly throughout the country, affecting tens of thousands of patients, including several thousands have requested hospitalization and some hospitalization in intensive care, putting a strain on the entire regional health system.

Patients that present intermediate severity of the infection are often treated with non-invasive ventilatory support which includes high-flow nasal cannulas (HFNC), non-invasive ventilation (NIV), continuous positive airway pressure (CPAP) through face mask or helmet (helmet).

The exponential growth in the number of patients has made the massive use of these devices necessary even outside the intensive or semi-intensive wards where they are traditionally used.

Epidemiological knowledge regarding the type of patients treated with this strategy and the outcome of these patients are limited, but very important in a context of emergency.

Thus, the objective of this prospective multicenter study is to evaluate the number of patients with COVID-19 related pneumonia, treated with non-invasive ventilatory support outside the intensive care unit and to evaluate the clinical characteristics and hospital outcomes of these patients.

SAMPLE SIZE (n. Patients):

The study will collect all patients with the inclusion criteria, so the study size being by definition equal to the maximum size.

STUDY DESIGN:

Patients will be enrolled on a single day (March 26, 2020 or March 31, 2020 chosen by the participating centres).

Total duration of the Study: 5 months (enrollment, collection and analysis of data).

Enrollment Start: March 26, 2020. Enrollment Closure: March 31, 2020. End of the Study (indicative date, last visit, last patient): May 2020.

The patient will be enrolled in the study when informed consent is obtained.

In this phase, the following data are collected:

* Patient registration;
* Demographic and anthropometric data;
* Comorbidity
* Hospitalization data;
* Ventilation / Hemodynamics data;
* Blood chemistry tests.

Upon discharge other data will be collected such as the necessary intubation or intubation date.

STATISTICAL ANALYSIS:

The enrolled cases will be counted and the percentages of the three types of non-invasive ventilatory supports will be specifically described by centre. The heterogeneity of these percentages will be assessed through a model with mixed effects.

The anamnestic and clinical data of the enrolled patients will be analysed through descriptive statistics on continuous quantitative variables.

The impact of the type of ventilation and of the blood chemistry parameters and aspects of comorbidity will be assessed with reference to the probability of developing a transition to the death and to hospitalization in intensive care through a multinomial model.

These factors will also be included in a logistic model with outcome defined by patient survival.

ELIGIBILITY:
Inclusion Criteria:

* Age> = 18 years
* Diagnosis of COVID-related pneumonia requiring non-invasive ventilatory support (high-flow nasal cannula, and / or non-invasive ventilation and / or CPAP)

Exclusion Criteria:

- Explicit refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted on all patients diagnosed with COVID-related pneumonia in need of non-invasive ventilatory support. Patients will be enrolled on single day (March 26, 2020 or March 31, 2020 chosen by the participating centers).
Sampling Method: Non-Probability Sample
Enrollment: 909 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
The number of patients treated with non-invasive ventilation devices. | Until patient discharge from the hospital (approximately 5 months)
  The first purpose of the study is to evaluate the number of COVID-19 related pneumonia patients treated with devices for non-invasive ventilation outside intensive care units.

SECONDARY OUTCOMES:
Incidence of patients requiring mechanical ventilation | Until patient discharge from the hospital (approximately 5 months)
  Assess the clinical characteristics of patients treated with devices for non-invasive ventilation using the following endpoint: incidence of patients requiring mechanical ventilation.
Incidence of organ failure | Until patient discharge from the hospital (approximately 5 months)
  Assess the clinical characteristics of patients treated with devices for non-invasive ventilation using the following endpoint: incidence of organ failure.
Duration of hospitalization | Until patient discharge from the hospital (approximately 5 months)
  Measure the hospital outcomes of patients treated with devices for non-invasive ventilation using the following endpoint: duration of hospitalization.
Clinical outcome at hospital discharge | Until patient discharge from the hospital (approximately 5 months)
  Measure the hospital outcomes of patients treated with devices for non-invasive ventilation using the following endpoint: clinical outcome at hospital discharge.

CONTACTS AND LOCATIONS:
Locations (34):
- Italy (34):
  - Policlinico San Marco - Ospedale Zingonia, Bergamo, BG
  - ASST Papa Giovanni XXIII - Bergamo, Bergamo
  - Azienda Ospedaliera - Universitaria di Bologna, Policlinico S. Orsola Malpighi, Bologna
  - ASST Spedali Civili - Brescia, Brescia
  - ASST Valle Olona - Ospedale di Busto Arsizio, Busto Arsizio
  - ASST Lariana - Ospedale Sant'Anna, Como
  - ASST Crema - Ospedale Maggiore di Crema, Crema
  - ASST Cremona - Ospedale di Cremona, Cremona
  - Istituto Clinico Humanitas Gavazzeni, Cremona
  - ASST Garda - Presidio di Desenzano del Garda, Desenzano del Garda
  - ASST Monza - Desio, Desio
  - ASST Spedali Civili -Ospedale di Gardone Val Trompia, Gardone Val Trompia
  - ASST Lecco - Ospedale "A. Manzoni", Lecco
  - ASST Ovest milanese - Ospedale di Legnano, Legnano
  - ASST Lodi - Ospedale Maggiore di Lodi, Lodi
  - ASST OVEST Milanese - Ospedale di Magenta, Magenta
  - ASST Garda - Ospedale di Manerbio, Manerbio
  - ASST Mantova - Ospedale Carlo Poma, Mantova
  - ASST Melegnano e della Martesana - Presidio di Melzo-Gorgonzola, Melzo
  - ASST Fatebenefratelli - Presidi Fatebenefratelli & M. Melloni, Milan
  - ASST Fatebenefratelli - Sacco, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Giuseppe, Milan
  - ASST Spedali Civili -Presidio Ospedaliero di Montichiari, Montichiari
  - ASST Monza - Ospedale San Gerardo, Monza
  - Fondazione IRCCS Policlinico San Matteo - Pavia, Pavia
  - Policlinico San Pietro, Ponte San Pietro
  - Istituto Clinico Humanitas Rozzano, Rozzano
  - ASST Valle Olona - Ospedale di Saronno, Saronno
  - ASST Bergamo OVEST - Ospedale "Treviglio-Caravaggio" di Treviglio, Treviglio
  - Ospedale di Circolo e Fondazione Macchi - Varese, Varese
  - ASST Vimercate - Ospedale di Vimercate, Vimercate
  - ASST Melegnano e della Martesana - Ospedale di Vizzolo Predabissi, Vizzolo Predabissi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Derived] Bellani G, Grasselli G, Cecconi M, Antolini L, Borelli M, De Giacomi F, Bosio G, Latronico N, Filippini M, Gemma M, Giannotti C, Antonini B, Petrucci N, Zerbi SM, Maniglia P, Castelli GP, Marino G, Subert M, Citerio G, Radrizzani D, Mediani TS, Lorini FL, Russo FM, Faletti A, Beindorf A, Covello RD, Greco S, Bizzarri MM, Ristagno G, Mojoli F, Pradella A, Severgnini P, Da Macalle M, Albertin A, Ranieri VM, Rezoagli E, Vitale G, Magliocca A, Cappelleri G, Docci M, Aliberti S, Serra F, Rossi E, Valsecchi MG, Pesenti A, Foti G. Noninvasive Ventilatory Support of Patients with COVID-19 outside the Intensive Care Units (WARd-COVID). Ann Am Thorac Soc. 2021 Jun;18(6):1020-1026. doi: 10.1513/AnnalsATS.202008-1080OC. PMID 33395553